CLINICAL TRIAL: NCT03904290
Title: Does Patent Foramen Ovale Closure Improve Exercise Capacity & Prevent Blood Flow Through Intrapulmonary Shunt
Acronym: PFO CLOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12132016.027
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Intervention Model Description: Subjects brought in for testing prior to PFO closure, then testing repeated 3 months post PFO closure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-PFO closure (Other): Subjects evaluated at 'baseline' prior to percutaneous closure of PFO, and re-evaluated at 3 months post percutaneous closure of PFO
  Interventions: Other: PFO Closure

INTERVENTIONS:
Other: PFO Closure — Subject will undergo percutaneous closure of PFO/ASD utilizing FDA-approved PFO/ASD closure device(s).

SUMMARY:
The overarching goal of this study is to examine cardiopulmonary and respiratory physiology pre and post PFO/ASD closure in patients who are undergoing surgical closure of their PFO/ASD.

DETAILED DESCRIPTION:
A patent foramen ovale (PFO) is present in ~30% of the general population. The PFO has historically been considered to be trivial. However, recent work by the investigator's group and others has identified that, compared to individuals without a PFO, those with a PFO have a higher core body temperature, significantly worse pulmonary gas exchange efficiency, blunted ventilatory responses to chronic hypoxia and acute carbon dioxide and increased susceptibility to altitude illnesses such as acute mountain sickness, and high altitude pulmonary edema. Specific to this application, subjects with a PFO maybe worse pulmonary gas exchange efficiency because a PFO is a potential source of right-to-left shunt that will make pulmonary gas exchange efficiency worse. If true, then this may negatively impact exercise capacity and/or exercise tolerance.

The investigator's lab group has demonstrated that hypoxemia increases blood flow through intrapulmonary arteriovenous anastomoses (IPAVA) in healthy and subjects with COPD. When these subjects breathe 100% O2 it prevents or reduces blood flow through IPAVA. This suggests that hypoxemia per se induces blood flow through IPAVA. The blood flow through IPAVA and presence of a PFO is also associated with increased risk of stroke and/or transient ischemic attack (TIA). In addition, an atrial septal defect (ASD) is a hole within the interatrial septum, and is considered a congenital heart defect. An ASD is typically larger than a PFO, and thus, the symptoms may be worse in those with an ASD, compared to those with a PFO. Thus, some hypoxemic patients who have had a stroke or transient ischemic attack, who also have a PFO/ASD may undergo surgical closure of their PFO/ASD to prevent subsequent neurological sequelae. This surgical closure may also prevent the hypoxemia thereby reducing or preventing blood flow through IPAVA. Of note, blood flow through IPAVA has been demonstrated to be strongly correlated with TIA and/or stroke and has not previously been taken into consideration in randomized clinical trials mentioned below.

Three randomized clinical trials have determined that PFO closure is not superior to regular medical management, for the prevention of subsequent stroke and/or TIA. Nevertheless, the American Heart Association still recommends that "in patients with cryptogenic [unexplained] TIA or stroke, a PFO, and deep vein thrombosis (DVT), guidelines from the American College of Chest Physicians currently recommend vitamin K antagonist therapy for 3 months and consideration of PFO closure rather than no vitamin K antagonist therapy or aspirin therapy." Additionally, in the largest single center retrospective study performed to date, PFO closure for the purpose of preventing hypoxemia was found to result in "improvement in echocardiographic evidence of right to left shunt, New York Heart Association functional class, and oxygen requirement." Thus, PFO/ASD closure remains a potentially beneficial option for both hypoxemic and stroke/TIA patients.

Lastly, preliminary data also suggest greater levels of plasma inflammatory mediators in subjects with a PFO and systemic inflammation is associated with increased risk of cardiovascular diseases. Importantly, exercise is known to reduce so of these systemic inflammatory mediator levels. Thus, PFO/ASD closure may allow for greater exercise capacity and a subsequent reduction in inflammation.

Thus, although a PFO has been traditionally considered to have a minimal impact of physiology and pathophysiology, emerging evidence suggests this may not be the case. The investigator's lab is focused on understanding how and why a relatively small hole in the heart (PFO/ASD) can have a relatively large impact on cardiopulmonary and respiratory physiology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-80
* Undergoing PFO/ASD closure.
* Subject's physician will determine inclusion in either exercise or non-exercise group, based on available medical information.

Exclusion Criteria:

* Previous history of coronary artery disease (ischemic heart disease such as angina, heart attack, myocardial infarction).
* Failure of Modified Allen's Test in both hands.
* Currently taking medications or herbal supplements for any heart or respiratory disease that they cannot stop taking for 48hrs prior to testing (seasonal allergy medication not included in exclusion medications).
* Lidocaine, nitroglycerine or heparin allergy.
* Women who are pregnant or trying to become pregnant.
* Previous history of any condition that would prevent the subject from performing cycle ergometer exercise (for exercise study only).
* Physician determination.
* PFO/ASD deemed by referring physician as not fully closed/endothelialized at 6 months post-PFO/ASD closure procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quantified pulmonary gas exchange efficiency | Baseline and 3 months post percutaneous closure
  Quantify pulmonary gas exchange efficiency (alveolar to arterial O2 difference) and arterial oxygenation at rest and during exercise.
change in maximal aerobic exercise capacity (Vo2max) | Baseline and 3 months post percutaneous closure
  Quantify aerobic exercise capacity as measured by oxygen consumption
change in maximal aerobic exercise capacity | Baseline and 3 months post percutaneous closure
  Distance walked in 6 minutes (6 minute walk test)
Change in minute flow of intrapulmonary arterio-venuous anastamoses (QIPAVA) | Baseline and 3 months post percutaneous closure
  Quantify QIPAVA at rest and assess recurrence of stroke or TIA at 3 months.
Change in plasma inflammatory markers | Baseline and 3 months post percutaneous closure
  Quantify plasma inflammatory markers (TNFa, IL-1, 6 & CRP)
Change in hypercapnic ventilatory response | Baseline and 3 months post percutaneous closure
  Measure hypercapnic ventilatory response
change in core body temperature measured via ingestible thermometer pill | Baseline and 3 months post percutaneous closure
  Quantify core body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lovering, PhD, Principal Investigator — University of Oregon
Locations (1):
- Cardiorespiratory and Pulmonary Physiology Lab, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03904290/Prot_SAP_000.pdf